CLINICAL TRIAL: NCT00119691
Title: Nesiritide Infusion for the Treatment of Decompensated Heart Failure and Renal Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Principal Investigator, Anju Nohria, Associate Physician/Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-P00235
Record Dates: First submitted 2005-07-07; First posted 2005-07-14 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Congestive Heart Failure; Renal Insufficiency
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nesiritide + standard of care (Experimental): Nesiritide: 1 mcg/kg bolus, followed by a continuous infusion at 0.005 mcg/kg/min which can be titrated every 3 hours by 0.005 mcg/kg/min to maximum dose of 0.03 mcg/kg/min until adequate diuresis achieved.
  Interventions: Drug: Nesiritide
- Standard of care (Active Comparator): Standard of care until adequate diuresis achieved
  Interventions: Drug: Nesiritide

INTERVENTIONS:
Drug: Nesiritide — Nesiritide: 1 mcg/kg bolus, followed by a continuous infusion at 0.005 mcg/kg/min which can be titrated every 3 hours by 0.005 mcg/kg/min to maximum dose of 0.03 mcg/kg/min until adequate diuresis achieved.
  Other Names: Natrecor

SUMMARY:
The researchers hypothesize that the addition of nesiritide to standard therapy will prevent worsening of renal function in patients admitted to the hospital with decompensated heart failure and renal dysfunction relative to standard therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated heart failure hospitalization with at least 1 symptom and 1 sign of elevated filling pressures
* Admission estimated creatinine clearance =< 50 cc/min.

Exclusion Criteria:

* Systolic blood pressure < 85 mm Hg
* Cardiogenic shock
* Volume depletion
* Myocardial infarction, unstable angina within last 30 days
* Significant valvular stenosis, hypertrophic/restrictive cardiomyopathy, or constrictive pericarditis
* Chronic hemodialysis
* Anticipated major procedure during hospitalization i.e. left heart catheterization, surgery, or transplantation
* Enrolled in another research protocol within last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Renal function | within 7 days after randomization

SECONDARY OUTCOMES:
Weight loss | Within 7 days from randomization
Days to optimal volume status | From randomization till day 7 or sooner
Concomitant diuretic use | Within 7 days from randomization
Global symptom assessment | 24 hrs and 3 days after randomization
Length of stay | From admission to discharge or day 7

CONTACTS AND LOCATIONS:
Overall Officials: Anju Nohria, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States